CLINICAL TRIAL: NCT04006990
Title: The Bed Rest Avoidance Study
Acronym: BRAVE
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Southern California (Other)
Collaborators: University of California, Los Angeles (Other)
Responsible Party: Principal Investigator, Brad Spellberg, Professor & Associate Dean, University of Southern California
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: HS-16-00804
Record Dates: First submitted 2019-07-01; First posted 2019-07-05 (Actual); Last update posted 2023-11-08 (Actual); Status verified 2023-11

CONDITIONS: Study Focuses on Bed Rest and Deconditioning in Hospital Inpatients

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Subjects are given recliner chairs and education on the dangers of bedrest
  Interventions: Behavioral: Provision of recliner chairs and encouragement to get out of bed
- Control (No Intervention): Subjects are treated with standard care

INTERVENTIONS:
Behavioral: Provision of recliner chairs and encouragement to get out of bed — Provision of recliner chairs and encouragement to get out of bed
  Arms: Intervention

SUMMARY:
Hospitalized patients spend the majority of their time lying in bed, even when they are capable of being out of bed. Up to 50% of inpatients suffer functional decline at least in part due to lying in bed after admission, and even those who are not placed on bed rest by their physicians spend an average of 20 out of 24 hours lying in bed. The loss of functional ability and exercise tolerance happens remarkably fast, as early as hospital day 2 (24-48 hours). Functional decline often results in a prolonged hospital stay and the need for additional rehabilitation resources both during and after the hospitalization to return a patient to their baseline functional status. Functional decline has also been associated with excess mortality.

The investigators sought to flip the culture of hospital-based care such that the bed was viewed as a place for patients to sleep, and patients would be encouraged to get out of bed when they were not trying to sleep. The investigators hypothesized that patients were unaware of the risks of prolonged immobilization and that the lack of an alternative comfortable place for patients to sit other than their bed contributed to their immobility. Previous studies have demonstrated that mobility protocols improve patient-centered outcomes in narrow patient populations such as post-surgical patients or the elderly, but such interventions have not been studied in a heterogeneous patient population. Additionally, previously studied protocols have been labor-intensive from a nursing standpoint, requiring, for example, that staff provide one-on-one supervised ambulation 3-4 times per day. The investigators aimed to determine whether establishing a relatively low-intensity, pragmatic protocol to discourage patients from lying in bed would result in shorter length of stay by improving mobility. The investigators further aimed to assess the additional impact of providing a recliner chair, a safe and comfortable alternative to their bed on these outcomes.

This a prospective, controlled investigation of a novel intervention intended to reduce time subjects spent lying in bed. The intervention will be conducted at Los Angeles County + University of Southern California (LAC+USC) Medical Center from March 20, 2017 through September 19, 2017. The intervention and control wards are symmetrically laid out. All wards consist of medical/surgical beds without cardiac telemetry monitoring. Subjects will be admitted per clinical routine, with bed assignments made by the bed control department, which was not aware of the study. Handouts developed at a 3rd grade level will inform subjects and their families about the risks of bed rest and encouraged the subjects to only lie in bed when they were attempting to sleep. Handouts are translated into 5 languages (Spanish, Korean, Tagalog, Mandarin, Vietnamese). Nursing staff on the intervention wards will provide these handouts to subjects and their families as part of the standard admission process. In addition, laminated reminder signs identical to the handouts will be posted on the wall opposite the head of the bed. Posters were placed in the main entrance of the study units.

Half of the intervention rooms will also be provided with recliner chairs (Winco Vero Care Cliner) that were bariatrics rated to 500 pounds, vinyl-covered for facile disinfection, and had 180-degree swing arms and locking casters. The other intervention rooms and the control rooms had standard hospital chairs in addition to the hospital bed.

The primary outcome measure is the difference in the length of hospital stay for admissions to intervention rooms compared to control rooms. Subjects' age and gender will be collected in order to control for these factors in the primary analysis. The Medicare Severity Diagnosis Related Group (MS DRG) relative weight for each patient will be collected to control for illness severity.

As a secondary endpoint, functional status will be assessed using the "6-Clicks" objective functional scoring system. Scores will be measured at several points during the each hospitalization As a process measure, nurses will maintain a log of hours per shift that subjects spend in bed. Finally, as a safety measure, the rates of falls per 1000 patient-days will be collected.

Data will be abstracted using an automated query of the electronic health record's bed management database (Cerner, Kansas City, MO). All patients who are placed on one of the study wards during the intervention period-including those admitted from the emergency department, elective medical and surgical admissions, inter-hospital transfers and intra-hospital transfers-will be included.

ELIGIBILITY:
Inclusion Criteria:

* Hospital Inpatient
* Admitted to the LAC+USC study wards during the study period

Exclusion Criteria:

* Age < 18

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6089 (Actual)
Dates: Start 2017-03-20 (Actual); Primary Completion 2017-09-19 (Actual); Study Completion 2017-09-19 (Actual)

PRIMARY OUTCOMES:
Hospital Length of Stay | 1 year

SECONDARY OUTCOMES:
Six Clicks Functional Score | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Brad Spellberg, MD, Principal Investigator — LAC+USC Medical Center
Locations (1):
- LAC USC Medical Center, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No